CLINICAL TRIAL: NCT06030479
Title: Topical Adrenaline Versus Warm Saline Solution for Minimizing Intraperitoneal Bleeding During Caesarian Delivery for Placenta Previa / Accreta Spectrum ( PAS): A Randomized Controlled Study
Brief Title: Topical Adrenaline Versus Warm Saline Solution for Minimizing Intraperitoneal Bleeding During Caesarian Delivery for Placenta Previa / Accreta Spectrum ( PAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MS-469-2023
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Placenta Accreta; Placenta Previa
MeSH Terms: conditions — Placenta Accreta; Placenta Previa | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Adrenaline Group (Experimental): Topical adrenaline group
  Interventions: Drug: Topical adrenaline
- Warm saline Group (Placebo Comparator): Warm saline Group
  Interventions: Drug: Warm saline

INTERVENTIONS:
Drug: Topical adrenaline — Skin is incised midline sub-umbilical incision , bladder dissection will be done , uterus will be incised by vertical upper segment incision , followed by delivery of the baby.
  Surgical assessment and decision for either conservative management or CS hysterectomy will be done.
  After completion of surgical procedure , surgical field is observed for major bleeding and patients are subjected to intervention Packing the pelvic surgical field with towels fully saturated with adrenaline 1:10000 solution.
  Arms: Topical Adrenaline Group
Drug: Warm saline — Skin is incised midline sub-umbilical incision , bladder dissection will be done , uterus will be incised by vertical upper segment incision , followed by delivery of the baby.
  Surgical assessment and decision for either conservative management or CS hysterectomy will be done.
  After completion of surgical procedure , surgical field is observed for major bleeding and patients are subjected to intervention Packing the surgical field with towels fully saturated with warm saline solution ( 50 degrees).
  Arms: Warm saline Group

SUMMARY:
Placenta accreta spectrum (PAS), encompassing the terms placenta accreta, increta, and percreta; abnormally invasive placenta; morbidly adherent placenta; and invasive placentation, is a leading cause of life-threatening obstetric haemorrage . Currently, more than 90% of women diagnosed with PAS also have a placenta praevia , and the combination of both conditions leads to high maternal morbidity and mortality due to massive haemorrhage at the time of birth . Maternal mortality of placenta praevia with percreta has been reported to be as high as 7% of cases .

Adrenaline has also been demonstrated to be a reasonable hemostatic agent because of its low cost, low risk, powerful vasoconstrictor, and platelet aggregation. Topical use of adrenaline is an effective and reasonable hemostatic agent in tonsillectomy.

DETAILED DESCRIPTION:
* Population of study: A total of 84 pregnant patients with placenta previa / Accreta spectrum.
* Study location: Obstetrics and Gynecology Kasr Al-Ainy Hospital , Faculty of Medicine , Cairo University.

This is a randomized controlled trial including a total number of 84 patients representing study group , randomized in 2 equal groups , using computer generated randomization sheet on (Medcalc ®) .

Group A : Topical adrenaline group (n=42)

Group B : Warm saline Group (control) (n=42)

The aim of the study is to evaluate the efficacy of topical adrenaline for decreasing intraperitoneal bleeding during caesarian section for placenta previa/ Accreta spectrum (PAS).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 40 years.
* BMI < 35.
* Pregnant patients with placenta previa .
* Placenta accrete spectrum.
* Vitally stable .

Exclusion Criteria:

* Vitally unstable .
* Massive pre- or intra-operative bleeding.
* Medical disorders ( e.g. : hypertension , cardiac …. )

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
control of intra-operative bleeding from surgical field. | 30 minutes after application of topical drug
  control of intra-operative bleeding from surgical field if bleeding stopped , or minimal oozing , towel are not soaked with blood and improvement of general condition with no hemoglobin drop.

SECONDARY OUTCOMES:
Need for hemostatic sutures , uterine artery ligation , internal iliac artery ligation , hysterectomy | if bleeding continued 30 minutes after topical drugs
  Need for hemostatic sutures , uterine artery ligation , internal iliac artery ligation , hysterectomy
immediate maternal complications ( postpartum haemorrage , DIC , hysterectomy , maternal mortality , ICU admission , …) | 24 hours after delivery
  immediate maternal complications ( postpartum haemorrage , DIC , hysterectomy , maternal mortality , ICU admission , …)

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Solheim KN, Esakoff TF, Little SE, Cheng YW, Sparks TN, Caughey AB. The effect of cesarean delivery rates on the future incidence of placenta previa, placenta accreta, and maternal mortality. J Matern Fetal Neonatal Med. 2011 Nov;24(11):1341-6. doi: 10.3109/14767058.2011.553695. Epub 2011 Mar 7. PMID 21381881
- [Background] Jauniaux E, Bhide A, Kennedy A, Woodward P, Hubinont C, Collins S; FIGO Placenta Accreta Diagnosis and Management Expert Consensus Panel. FIGO consensus guidelines on placenta accreta spectrum disorders: Prenatal diagnosis and screening. Int J Gynaecol Obstet. 2018 Mar;140(3):274-280. doi: 10.1002/ijgo.12408. No abstract available. PMID 29405319
- [Background] Hatton RC. Bismuth subgallate-epinephrine paste in adenotonsillectomies. Ann Pharmacother. 2000 Apr;34(4):522-5. doi: 10.1345/aph.19216. PMID 10772440